CLINICAL TRIAL: NCT04099043
Title: Cascade Continuous Glucose Monitor 15-day Performance Assessment
Brief Title: Cascade CGM 15-day Performance Assessment
Acronym: CASPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WaveForm Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR-19-0032
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-09

CONDITIONS: Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Monitoring (Experimental): Single Arm, Randomized
  Interventions: Device: Cascade Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Cascade Continuous Glucose Monitoring System — Continuous Glucose Monitoring for 15 days

SUMMARY:
To validate the feasibility of a 15-day wear period of the Cascade CGM system

DETAILED DESCRIPTION:
To assess a 15-day wear period for the Cascade CGM. This study includes ten subjects who will interface with the system and take finger stick BGM glucose values for calibration. The wear period includes four in-clinic days frequent blood draws and eleven at home days at a single testing site.

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent form

  * Diagnosis of type 1 or type 2 (on insulin therapy) diabetes mellitus for at least 6 months
  * 18 years of age or older
  * Currently self-monitoring capillary blood glucose (on average at least three times per day or more) or on a CGM for at least three months
  * Willing to have blood glucose levels manipulated into high and low glucose levels during in clinic days if deemed appropriate per the protocol based on insulin use.
  * Willing to follow all study procedures, including attending all clinic visits during which a venous line will be inserted for blood sampling, wearing CGM sensors for entire study, performing fingertip glucose tests for self-monitoring and calibration, and keeping a diary of activities.
  * Be willing to wear two investigational CGM devices.

Exclusion Criteria:

* • Known allergy to medical grade adhesives

  * Magnetic Resonance Imaging (MRI) scheduled during CGM sensor wear period
  * Persons with type 2 diabetes using diet and exercise only for diabetes management
  * Used an investigational drug within 30 days prior to study entry
  * Hematocrit < 32% (obtained during screening)
  * Inadequate veins (in the opinion of the investigator) or known contraindication to placement of a dedicated peripheral line for venous blood withdrawal
  * Symptomatic coronary artery disease with a history of angina, or history of a myocardial infarction or coronary intervention (e.g., percutaneous transluminal coronary angioplasty [PTCA], stent placement), or coronary artery bypass graft (CABG) within the past six months
  * Diagnosis of the following diabetic autonomic neuropathies: orthostatic hypotension, heart rate anomalies, gastroparesis
  * Cerebrovascular incident within the past six month
  * History or presence of eczema, psoriasis, atopic or contact dermatitis
  * Subject is pregnant at the start of the study.
  * Current use or within one-week exposure to topical medications at the proposed insertion sites
  * Seizure disorder (epilepsy)
  * Malignancy within the past five years, except basal cell or squamous cell skin cancers
  * Major surgical operation within 30 days prior to screening
  * Other medical conditions that would pose safety concerns, interfere with study conduct or seriously compromise study integrity (reason for exclusion will be clearly documented by investigator or designee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-28 (Actual); Primary Completion 2019-10-13 (Actual); Study Completion 2019-10-13 (Actual)

PRIMARY OUTCOMES:
15-day Continuous Glucose Monitoring | Fifteen days
  Fifteen days of sensor wear with the Cascade CGM Smart Device App

CONTACTS AND LOCATIONS:
Overall Officials: Maja Navodnik Peložnik, MD, Principal Investigator — Splošna bolnišnica Celje
Locations (1):
- Splošna bolnišnica Celje, Celje, Slovenia

IPD SHARING:
Plan to Share IPD: No